CLINICAL TRIAL: NCT06220253
Title: Comparison of Learning Curves for Two Different Techniques in Vaginal Hysterectomy: Traditional Versus Minimally Invasive Bipolar Coagulation Technique
Brief Title: Comparison of Learning Curves for Two Different Techniques in Vaginal Hysterectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Salvatore, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LEACURV
Record Dates: First submitted 2022-06-06; First posted 2024-01-23 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse; Gynecologic Disorders; Surgery
Keywords: pelvic organ prolapse; urogynecologic surgery; learning curve; bipolar vessels sealing
MeSH Terms: conditions — Pelvic Organ Prolapse; Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 in two groups:
  1. Study group: bipolar coagulation technique
  2. Comparison group: reabsorbable stitches
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Hysterectomy by bipolar coagulation technique (Other): The surgery will take place according to the canonical times of vaginal hysterectomy, after incision of the portio, detachment of the bladder-vaginal fascia and vaginal rectum, opening of the anterior and posterior peritoneum, taking, section and ligament of the ligaments uterus-sacral ligaments, and subsequent coagulation by bipolar instrument of the other structures of the uterus and their section, in particular of the uterine arteries, tubes, uterine-ovarian ligaments and round ligament bilaterally.
  Interventions: Procedure: vaginal hysterectomy by bipolar vessels sealing
- Vaginal hysterectomy by traditional technique with reabsorbable stitches (Other): The surgery will take place according to the canonical times of vaginal hysterectomy, after incision of the port, detachment of the bladder-vaginal fascia and vaginal rectum, opening of the anterior and posterior peritoneum, taking and suturing with absorbable threads of all the support structures of the uterus, in particular uterus-sacral ligaments, uterine arteries, tubes, uterine-ovarian ligaments and round ligament bilaterally.
  Interventions: Procedure: vaginal hysterectomy by traditional technique

INTERVENTIONS:
Procedure: vaginal hysterectomy by bipolar vessels sealing — The surgery will take place according to the canonical times of vaginal hysterectomy and all the support structures will be coagulated and cut by a bipolar vessel sealing instrument
  Arms: Vaginal Hysterectomy by bipolar coagulation technique
Procedure: vaginal hysterectomy by traditional technique — The surgery will take place according to the canonical times of vaginal hysterectomy and all the support structures will be sutured by absorbable threads
  Arms: Vaginal hysterectomy by traditional technique with reabsorbable stitches

SUMMARY:
Randomized prospective monocentric interventional study to compare learning curves for traditional vaginal hysterectomy and vaginal hysterectomy performed by bipolar coagulation comparing short-term outcomes for both procedures.

DETAILED DESCRIPTION:
This is a prospective, randomized, spontaneous monocentric interventional study on a procedure in which 60 female patients will be enrolled with a diagnosis of pelvic organs prolapse which are eligible for vaginal hysterectomy. The data relating to the intervention will be collected, analyzed and compared through a descriptive statistics.

Patients will be randomized 1:1 in two groups:

1. Study group: bipolar coagulation technique
2. Comparison group: reabsorbable stitches The primary outcome of the study is to compare the learning curves for two vaginal surgical techniques for hysterectomy performed for the treatment of prolapse of the pelvic organs in women.

Secondary outcomes are to evaluate the effectiveness of the two different procedures through the evaluation of short-term outcomes for both procedures under consideration.

The planned duration of recruitment will be 7 months. In this period of time it is planned to enrol a total of 60 patients. Once the learning curve plateau has been reached for both procedures, the study will be considered finished. The number of samples was chosen on the basis of the feasibility of recruitment and the possibility of evaluating the learning curve of the operators.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >18 years
* Genital prolapse > II degree in accordance with the "POP-Q System" eligible for vaginal hysterectomy
* Understanding and signing of informed consent for surgical procedure

Exclusion Criteria:

* Need for simultaneous bilateral adnexectomy
* Previous cesarian section
* Patients with abdominal laparoscopic or laparotomy history
* Patients with malignant pathology and/or adnexal pathology
* Confirmed or presumed pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Learning curve comparison | immediate post operative time
  The primary objective of the study is to compare the learning curves (in terms of operating time, blood loss, intraoperative complications) for two vaginal surgical techniques for hysterectomy performed for the treatment of prolapse of the pelvic organs in women. The two procedures compared will be the traditional technique performed by applying reabsorbable sutures and the bipolar coagulation technique.

SECONDARY OUTCOMES:
Evaluate the effectiveness of the two different techniques of vaginal hysterectomy. | 3 days after the surgical procedure
  Effectiveness will be assessed in terms of short-term outcomes such as:
  Intraoperative complications post-operative pain inpatient time Post-operative urinary infections vaginal infections, postoperative collected hematomas

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Salvatore, MD, Principal Investigator — San Raffaele Hospital, Milan
Locations (1):
- Arianna Casiraghi, Milan, Italy